CLINICAL TRIAL: NCT04944563
Title: Comparison of Segmentectomy Versus Lobectomy for Early-stage Non-small Cell Lung Cancer ≤ 2 cm in the Middle Third of the Lung Field: A Prospective and Multi-center RCT Study
Brief Title: Comparison of Segmentectomy Versus Lobectomy for Non-small Cell Lung Cancer ≤ 2 cm in the Middle Third of the Lung Field
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-SR-164
Record Dates: First submitted 2021-06-17; First posted 2021-06-29 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Lung Neoplasms; Surgery
Keywords: Non-small cell lung cancer; Segmentectomy; Lobectomy; the middle third of the lung field
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Mastectomy, Segmental; Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Segmentectomy (Experimental): Patients receive segmentectomy
  Interventions: Procedure: Segmentectomy
- Lobectomy (Active Comparator): Patients receive lobectomy
  Interventions: Procedure: Lobectomy

INTERVENTIONS:
Procedure: Segmentectomy — Patients receive segmentectomy
  Arms: Segmentectomy
Procedure: Lobectomy — Patients receive lobectomy
  Arms: Lobectomy

SUMMARY:
This study aims to investigate whether segmentectomy had non-inferiority long-term oncological effects (disease-free survival and overall survival) compared with lobectomy in the treatment of patients with early-stage non-small cell lung cancer ≤ 2 cm in the middle third of lung field.

DETAILED DESCRIPTION:
Nowadays, the role of segment resection in the treatment of non-small cell lung cancer ≤ 2 cm in the outer third of the lung field has been evaluated in multiple studies. Recently, professor Hisao Asamura released the long-term results of the JCOG0802 project in AATS 2021. Segmentectomy had a higher 5-year overall survival (94.3% vs. 91.1%) than lobectomy (P < 0.001) for non-small cell lung cancer ≤ 2 cm (CTR > 0.5) in the outer third of the lung field. However, a substantial portion of lung nodules was not located in the outer third, but the middle third of the lung field. Whether segmentectomy has non-inferiority long-term oncological effects compared to lobectomy for early-stage non-small cell lung cancer ≤ 2 cm in the middle third of lung field remains unclear. This randomized controlled trial study aims to investigate whether segmentectomy has non-inferiority long-term oncological effects compared to lobectomy for early-stage non-small cell lung cancer ≤ 2 cm in the middle third of the lung field.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18-75 years old;
2. 6 mm ≤ tumor size ≤ 20 mm;
3. 0.25 < CTR < 1;
4. Center of tumor located in the middle third of the lung field;
5. ECOG score of 0,1 or 2;
6. Lung function (FEV1 ≥ 1 L and ≥ 70%);
7. Both lung segmentectomy and lobectomy could achieve R0 resection;
8. No serious cardiopulmonary complications, and could withstand both lung segmentectomy and lobectomy;
9. No hilus pulmonis and mediastinal lymph node metastasis and no distant metastasis;
10. Single tumor nodule or the concomitant nodule < microinvasive tumor;
11. Written informed consent.

Exclusion Criteria:

1. The tumor nodule is located in right middle lobe;
2. A history of other malignancies in the last 5 years (exclusion of early-staged thyroid cancer);
3. Have received preoperative anti-tumor therapy, including prior chemotherapy, radiation therapy, target therapy and so on;
4. A serious mental illness;
5. Pregnant and lactating women;
6. Congestive heart failure, myocardial infarction, severe stenosis of coronary artery within recent 6 months;
7. With the history of cerebral infarction or cerebral hemorrhage within 6 months;
8. With the history of sustained systemic corticosteroid therapy within 1 month;
9. The predicted surgical margin is less than 2 cm or the maximum diameter of the tumor at the 3D-CTBA
10. Other unsuitable situations;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
5-year Disease-Free Survival | From date of the recruitment, assessed up to 60 months
  The time interval from randomization to the earliest onset of any of the following events: tumor local recurrence, distant metastasis, and mortality

SECONDARY OUTCOMES:
30-day Morbidity and mortality rates | From date of the recruitment, assessed up to 30 days
  The rates of complications and death related to treatment during perioperative period
Pulmonary function in the first year after surgery | From date of the 3rd, 6th, and 12th month after surgery
  The Forced expiratory volume in one second (FEV1) in liter
3-year Disease-Free-Survival | From date of the recruitment, assessed up to 36 months
  The time interval from randomization to the earliest onset of any of the following events: tumor local recurrence, distant metastasis, and mortality
5-year overall Survival | From date of the recruitment, assessed up to 60 months
  The time interval from randomization to death caused by any reason

CONTACTS AND LOCATIONS:
Overall Officials: Liang Chen, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altorki NK, Wang X, Wigle D, Gu L, Darling G, Ashrafi AS, Landrenau R, Miller D, Liberman M, Jones DR, Keenan R, Conti M, Wright G, Veit LJ, Ramalingam SS, Kamel M, Pass HI, Mitchell JD, Stinchcombe T, Vokes E, Kohman LJ. Perioperative mortality and morbidity after sublobar versus lobar resection for early-stage non-small-cell lung cancer: post-hoc analysis of an international, randomised, phase 3 trial (CALGB/Alliance 140503). Lancet Respir Med. 2018 Dec;6(12):915-924. doi: 10.1016/S2213-2600(18)30411-9. Epub 2018 Nov 12. PMID 30442588
- [Background] Nakamura K, Saji H, Nakajima R, Okada M, Asamura H, Shibata T, Nakamura S, Tada H, Tsuboi M. A phase III randomized trial of lobectomy versus limited resection for small-sized peripheral non-small cell lung cancer (JCOG0802/WJOG4607L). Jpn J Clin Oncol. 2010 Mar;40(3):271-4. doi: 10.1093/jjco/hyp156. Epub 2009 Nov 22. PMID 19933688
- [Background] Suzuki K, Saji H, Aokage K, Watanabe SI, Okada M, Mizusawa J, Nakajima R, Tsuboi M, Nakamura S, Nakamura K, Mitsudomi T, Asamura H; West Japan Oncology Group; Japan Clinical Oncology Group. Comparison of pulmonary segmentectomy and lobectomy: Safety results of a randomized trial. J Thorac Cardiovasc Surg. 2019 Sep;158(3):895-907. doi: 10.1016/j.jtcvs.2019.03.090. Epub 2019 Apr 9. PMID 31078312
- [Background] Wu WB, Xia Y, Pan XL, Wang J, He ZC, Xu J, Wen W, Xu XF, Zhu Q, Chen L. Three-dimensional navigation-guided thoracoscopic combined subsegmentectomy for intersegmental pulmonary nodules. Thorac Cancer. 2019 Jan;10(1):41-46. doi: 10.1111/1759-7714.12897. Epub 2018 Nov 3. PMID 30390378
- [Background] Tsutani Y, Miyata Y, Nakayama H, Okumura S, Adachi S, Yoshimura M, Okada M. Appropriate sublobar resection choice for ground glass opacity-dominant clinical stage IA lung adenocarcinoma: wedge resection or segmentectomy. Chest. 2014 Jan;145(1):66-71. doi: 10.1378/chest.13-1094. PMID 24551879
- [Background] Wu W, He Z, Xu J, Wen W, Wang J, Zhu Q, Chen L. Anatomical Pulmonary Sublobar Resection Based on Subsegment. Ann Thorac Surg. 2021 Jun;111(6):e447-e450. doi: 10.1016/j.athoracsur.2020.10.083. Epub 2021 Jan 30. PMID 33524360